CLINICAL TRIAL: NCT02245867
Title: Phase Ia/Ib Study of Chimeric Fibril-Reactive Monoclonal Antibody 11-1F4 in Patients With AL Amyloidosis
Brief Title: Study of Chimeric Fibril-Reactive Monoclonal Antibody 11-1F4 in Patients With AL Amyloidosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAEL101-101; FDA Grant R01FD005110 (Other Grant/Funding Number: FDA OOPD); AAAM5108 (Other: Columbia University)
Record Dates: First submitted 2014-09-15; First posted 2014-09-22 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: AL Amyloidosis
Keywords: AL Amyloidosis; Amyloid, Light Chain Amyloidosis; Relapse; Refractory
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase Ia (Experimental): Administration of Chimeric Fibril-Reactive Monoclonal Anti-body 11-1F4:
  A 1-patient cohort will be infused with 0.5 mg/m2 of Ch 11-1F4 and, if tolerated, the doses in the next patients will be increased to 5, 10, 50, 100, 250, and finally, 500 mg/m2. All individuals will be evaluated prior to treatment, after infusion weekly for four weeks, as well as at 8 weeks.
  Interventions: Drug: Chimeric Fibril-Reactive Monoclonal Anti-body 11-1F4
- Phase Ib (Experimental): Administration of Chimeric Fibril-Reactive Monoclonal Anti-body 11-1F4:
  Subjects will receive four weekly infusions of the monoclonal anti-body at Dose Level 1 (0.5 mg/m2). If tolerated, the doses in the next patients will be increased to 5, 10, 50, 100, 250, and finally, 500 mg/m2. When the highest tolerated dose is reached without toxicity in 2 patients, an additional 4 patients will be enrolled and infused at that dose. Escalation or de-escalation will continue until we have determined the highest dose level at which less than 2 patients experience toxicity. All individuals will be evaluated prior to each course of treatment, as well as at weeks 5, 8, and 12.
  Interventions: Drug: Chimeric Fibril-Reactive Monoclonal Anti-body 11-1F4

INTERVENTIONS:
Drug: Chimeric Fibril-Reactive Monoclonal Anti-body 11-1F4 — The antibody binds to the pathologic material and initiates a neutrophil/macrophage response
  Other Names: Ch mAb 11-1F4

SUMMARY:
The purpose of this study is to examine the tolerance, safety, pharmacokinetics, and possible clinical benefit of the good manufacturing practice (GMP)-grade amyloid fibril-reactive chimeric (Ch) IgG1 mAb 11-1F4 in patients with amyloid light-chain (AL) amyloidosis.

The phase 1a part will involve at least 3 patients and a maximum of 18 patients. The first patient will receive the starting dose of the antibody and, if tolerated, the following patients will each receive (if tolerated) progressively higher doses of the antibody. Patients in part 1a of the trial will receive only one infusion of the drug. Patients treated in the phase 1a part receive lower dosage which might not be effective.

Once the maximal tolerated dosage is established during the phase 1a part, the investigators will accrue patients to the phase 1b part of the trial. Patients will receive 4 infusions, once each week for 4 weeks. Patients who were treated in the part 1a of the trial and showed no toxicity can be also treated in the part 1b of the trial. The first patient will receive the starting dose of the antibody and, if tolerated, the following patients will each receive (if tolerated) progressively higher doses of the antibody. When the investigators reach the maximum tolerated dose without toxicity, the investigators will enroll another 4 patients to receive the same dose. If there are no toxicities, another 4 patients will be treated at the next dose level, and so forth. Patients treated in Phase 1b may receive lower dosages which might not be effective. The goal of Phase 1b is to establish the tolerance and possible beneficial effects of 11-1F4. If successful, treatment with this antibody would represent a novel approach in the care of individuals with AL amyloidosis.

DETAILED DESCRIPTION:
Presently, treatment of patients with amyloid light chain (AL) amyloidosis is limited to reducing production of the amyloid-forming light-chain protein by giving conventional or high-dose (with stem cell transplant) anti-plasma cell chemotherapy, as used for patients with multiple myeloma. Although this approach has extended survival, the prognosis remains poor due to the persistence or progression of the amyloid deposits in vital organs, such as the heart or kidney. A different treatment strategy would be to attempt to reduce and/or eliminate these deposits. This study evaluates this by administering an anti-amyloid monoclonal antibody, 11-1F4. This compound has been shown to reduce/destroy this material in an experimental animal model of amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of AL amyloidosis based on accepted clinical and laboratory criteria.
* Patients are greater than 21 years old.

  * Female patients are not of child bearing potential or if they are of child bearing potential, they must not be pregnant or breast-feeding.
  * Patients have a life expectancy greater than 3 months.
  * Patients have an Eastern Cooperative Oncology Group (ECOG)-specified performance status of less than or equal to 3.
* Patients to be included are those with measurable, localized amyloid deposits (larynx, subcutaneous tissue, muscle, lung, lymph nodes) or clinically evident systemic disease (liver, kidney, heart, etc).
* Only patients with prior systemic therapy with relapsed/refractory disease are eligible, unless they have declined or are not eligible for high-dose melphalan and autologous hematopoietic stem cell transplant (HSCT) or any other standard therapy that has been known to be life-prolonging or life-saving.
* Patients have adequate organ function.
* Patients with cancer are eligible provided they meet specific criteria.
* Patients must provide signed, written, informed consent and be willing and able to comply with eligibility requirements, scheduled, visits, and follow-up studies.

Exclusion Criteria:

* Non-AL amyloidosis.
* Renal failure (on dialysis).
* Females who are pregnant or breast-feeding.
* ECOG Performance Status greater than 3.
* Seriously limited cardiac, renal, or hepatic function.
* Uncontrolled infection or significant co-morbidity (e.g., uncontrolled diabetes, severe diarrhea).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Ch mAb 11-1F4 | 2 years approximately
  The MTD of a single application of Ch mAb 11-1F4 is defined as the highest safely-tolerated dose (mg/m2) where 0 patients experiences Dose Limiting Toxicity.

SECONDARY OUTCOMES:
Number of subjects with positive amyloid-related organ response | 12 weeks
  Amyloid-related organ response will be evaluated on the basis of the accepted criteria per consensus guidelines for the conduct and reporting of clinical trials in systemic light-chain amyloidosis, in patients who completed phase 1b.
Estimated mean area under the curve (AUC) for Ch mAb 11-1F4 | Phase 1a: 1, 2, 24 hours post start of infusion; then post-infusion week 1, 2, 3, 4, 8. Phase 1b: pretreatment, 1, 2, 24 hours post start of infusion; then post-infusion week 5, 8, 12.
  This is designed to determine the pharmacokinetics of Ch mAb 11-1F4 when given as a single intravenous (i.v.) infusion (phase 1a) or as a series of four weekly intravenous infusions (phase 1b).
Number of participants with adverse events | 2 years approximately
  This to obtain additional safety data of Ch mAb 11-1F4 when given as a single intravenous infusion (phase 1a) or as a series of four weekly intravenous infusions (phase 1b) by obtaining adverse event information for all subjects during active follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Eisenberger, MD, Principal Investigator — CUMC
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Solomon, A. and Weiss, D.T. Protein and host factors implicated in the pathogenesis of light chain amyloidosis (AL amyloidosis). Amyloid: Inter. J. Exper. Clin. Invest. 2: 269-279, 1995.
- [Background] Kyle RA, Gertz MA. Primary systemic amyloidosis: clinical and laboratory features in 474 cases. Semin Hematol. 1995 Jan;32(1):45-59. No abstract available. PMID 7878478
- [Background] Merlini G, Bellotti V. Molecular mechanisms of amyloidosis. N Engl J Med. 2003 Aug 7;349(6):583-96. doi: 10.1056/NEJMra023144. No abstract available. PMID 12904524
- [Background] Kyle RA, Gertz MA, Greipp PR, Witzig TE, Lust JA, Lacy MQ, Therneau TM. A trial of three regimens for primary amyloidosis: colchicine alone, melphalan and prednisone, and melphalan, prednisone, and colchicine. N Engl J Med. 1997 Apr 24;336(17):1202-7. doi: 10.1056/NEJM199704243361702. PMID 9110907
- [Background] Palladini G, Anesi E, Perfetti V, Obici L, Invernizzi R, Balduini C, Ascari E, Merlini G. A modified high-dose dexamethasone regimen for primary systemic (AL) amyloidosis. Br J Haematol. 2001 Jun;113(4):1044-6. doi: 10.1046/j.1365-2141.2001.02859.x. PMID 11442500
- [Background] Comenzo RL, Gertz MA. Autologous stem cell transplantation for primary systemic amyloidosis. Blood. 2002 Jun 15;99(12):4276-82. doi: 10.1182/blood.v99.12.4276. PMID 12036853
- [Background] Skinner M, Sanchorawala V, Seldin DC, Dember LM, Falk RH, Berk JL, Anderson JJ, O'Hara C, Finn KT, Libbey CA, Wiesman J, Quillen K, Swan N, Wright DG. High-dose melphalan and autologous stem-cell transplantation in patients with AL amyloidosis: an 8-year study. Ann Intern Med. 2004 Jan 20;140(2):85-93. doi: 10.7326/0003-4819-140-2-200401200-00008. PMID 14734330
- [Background] Landau H, Hassoun H, Rosenzweig MA, Maurer M, Liu J, Flombaum C, Bello C, Hoover E, Riedel E, Giralt S, Comenzo RL. Bortezomib and dexamethasone consolidation following risk-adapted melphalan and stem cell transplantation for patients with newly diagnosed light-chain amyloidosis. Leukemia. 2013 Apr;27(4):823-8. doi: 10.1038/leu.2012.274. Epub 2012 Sep 27. PMID 23014566
- [Background] O'Nuallain B, Allen A, Kennel SJ, Weiss DT, Solomon A, Wall JS. Localization of a conformational epitope common to non-native and fibrillar immunoglobulin light chains. Biochemistry. 2007 Feb 6;46(5):1240-7. doi: 10.1021/bi0616605. PMID 17260953
- [Background] O'Nuallain B, Allen A, Ataman D, Weiss DT, Solomon A, Wall JS. Phage display and peptide mapping of an immunoglobulin light chain fibril-related conformational epitope. Biochemistry. 2007 Nov 13;46(45):13049-58. doi: 10.1021/bi701255m. Epub 2007 Oct 18. PMID 17944486
- [Background] Hrncic R, Wall J, Wolfenbarger DA, Murphy CL, Schell M, Weiss DT, Solomon A. Antibody-mediated resolution of light chain-associated amyloid deposits. Am J Pathol. 2000 Oct;157(4):1239-46. doi: 10.1016/S0002-9440(10)64639-1. PMID 11021828
- [Background] Solomon A, Weiss DT, Wall JS. Immunotherapy in systemic primary (AL) amyloidosis using amyloid-reactive monoclonal antibodies. Cancer Biother Radiopharm. 2003 Dec;18(6):853-60. doi: 10.1089/108497803322702824. PMID 14969598
- [Background] Azeredo da Silveira S, Kikuchi S, Fossati-Jimack L, Moll T, Saito T, Verbeek JS, Botto M, Walport MJ, Carroll M, Izui S. Complement activation selectively potentiates the pathogenicity of the IgG2b and IgG3 isotypes of a high affinity anti-erythrocyte autoantibody. J Exp Med. 2002 Mar 18;195(6):665-72. doi: 10.1084/jem.20012024. PMID 11901193
- [Background] Wall J, Murphy CL, Solomon A. In vitro immunoglobulin light chain fibrillogenesis. Methods Enzymol. 1999;309:204-17. doi: 10.1016/s0076-6879(99)09016-3. PMID 10507026
- [Background] Solomon A, Weiss DT, Wall JS. Therapeutic potential of chimeric amyloid-reactive monoclonal antibody 11-1F4. Clin Cancer Res. 2003 Sep 1;9(10 Pt 2):3831S-8S. PMID 14506180
- [Background] Gertz MA, Comenzo R, Falk RH, Fermand JP, Hazenberg BP, Hawkins PN, Merlini G, Moreau P, Ronco P, Sanchorawala V, Sezer O, Solomon A, Grateau G. Definition of organ involvement and treatment response in immunoglobulin light chain amyloidosis (AL): a consensus opinion from the 10th International Symposium on Amyloid and Amyloidosis, Tours, France, 18-22 April 2004. Am J Hematol. 2005 Aug;79(4):319-28. doi: 10.1002/ajh.20381. PMID 16044444
- [Background] Davern S, Tang LX, Williams TK, Macy SD, Wall JS, Weiss DT, Solomon A. Immunodiagnostic capabilities of anti-free immunoglobulin light chain monoclonal antibodies. Am J Clin Pathol. 2008 Nov;130(5):702-11. doi: 10.1309/AJCPNS6K1CYJPDBA. PMID 18854262
- [Derived] Edwards CV, Rao N, Bhutani D, Mapara M, Radhakrishnan J, Shames S, Maurer MS, Leng S, Solomon A, Lentzsch S, Eisenberger A. Phase 1a/b study of monoclonal antibody CAEL-101 (11-1F4) in patients with AL amyloidosis. Blood. 2021 Dec 23;138(25):2632-2641. doi: 10.1182/blood.2020009039. PMID 34521113